CLINICAL TRIAL: NCT04038580
Title: A Comparative Assessment of Conventional and Adjustable Transfemoral Prosthetic Sockets
Brief Title: A Comparative Assessment of Transfemoral Prosthetic Sockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Deanna H Gates, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00140733
Record Dates: First submitted 2019-07-23; First posted 2019-07-31 (Actual); Results first posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Amputation; Amputation; Traumatic, Leg, Lower
Keywords: Socket; Transfemoral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Prescribed Laminated Socket (Sham Comparator): In this arm, participants will wear their clinically prescribed laminated socket. This period is approximately 2 weeks.
  Interventions: Device: Laminated Socket
- Adjustable Sockets (Experimental): In this condition, participants will be fitted with 3 different adjustable transfemoral sockets by a certified prosthetist. The order in which the sockets are fitted are randomized and the participant will spend approximately 4 weeks in each socket.
  Interventions: Device: Quatro; Device: Infinite Socket; Device: CJ Socket

INTERVENTIONS:
Device: Laminated Socket — This is the currently prescribed socket the participant normally wears.
  Arms: Prescribed Laminated Socket
Device: Quatro — The Quatro (Quorum) is one of three commercially available adjustable sockets used in this study that will be fit by a certified prosthetist.
  Arms: Adjustable Sockets
Device: Infinite Socket — The Infinite Socket (LiM Innovations) is one of three commercially available adjustable sockets used in this study that will be fit by a certified prosthetist.
  Arms: Adjustable Sockets
Device: CJ Socket — The CJ Socket (CJ Socket Technologies) is one of three commercially available adjustable sockets used in this study that will be fit by a certified prosthetist.
  Arms: Adjustable Sockets

SUMMARY:
The objective of the proposed work is to enhance understanding of the potential benefits of adjustable sockets and inform clinical decision making.

DETAILED DESCRIPTION:
The objective of the proposed work is to enhance understanding of the potential benefits of adjustable sockets and inform clinical decision making. The investigators will explore a range of outcomes that have been found to be important for prostheses users and specifically assess the claims made by device manufacturers. Thirty adults with a transfemoral amputation will participate in four test sessions; one with their clinically prescribed, laminated socket, and three with different adjustable sockets. This data will be used to test the following aims: 1) does socket design impact socket comfort and prosthetic satisfaction? 2) does socket design impact of prosthetic socket on patient mobility and confidence, 3) how does prosthetic socket design influences prosthetic use in the home?, and 4) Are individual characteristics associated with benefits of specific socket designs?

ELIGIBILITY:
Inclusion Criteria:

* Unilateral lower-limb amputation
* Six months of independent ambulation
* Own and regularly wear a prosthesis with socket
* Minimum functional level of K2 on the Medicare Functional Classification Level (MFCL): corresponding to "the ability or potential for ambulation with the ability to traverse low-level environmental barriers such as curbs, stairs, or uneven surfaces. Typical of the limited community ambulator"

Exclusion Criteria:

* Pathology or injury of the intact limb
* Medication that affects their ability to walk
* Neurologic or cardiovascular disease
* Significant vision problems
* Suffer from an impaired mental capacity that negatively impacts verbal communication with the clinicians and research team, or requires a Legally Authorized Representative to facilitate communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna H Gates, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Rosalind Franklin University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No
Participant data will be deidentified for publication.

RESULTS

PARTICIPANT FLOW:
Groups:
- Laminated, Then CJ, Then Infinite, Then Quatro; Laminated, Then CJ, Then Quatro, Then Infinite; Laminated, Then Infinite, Then CJ, Then Quatro; Laminated, Then Infinite, Then Quatro, Then CJ; Laminated, Then Quatro, Then Infinite, Then CJ; Laminated, Then Quatro, Then CJ, Then Infinite: Participants first complete testing with their prescribed prosthetic socket. Surveys were administered in the first visit, the participant completed functional testing, and then they wore wearable sensors for the subsequent week. They were then fit with each of three experimental sockets that they wore for a minimum of 4 weeks. Surveys were administered after three weeks and functional assessments occurred after 4 weeks. There was a 1-week washout between each condition.
Period: Baseline Testing
Arm/Group | Laminated, Then CJ, Then Infinite, Then Quatro | Laminated, Then CJ, Then Quatro, Then Infinite | Laminated, Then Infinite, Then CJ, Then Quatro | Laminated, Then Infinite, Then Quatro, Then CJ | Laminated, Then Quatro, Then Infinite, Then CJ | Laminated, Then Quatro, Then CJ, Then Infinite
Started | 5 | 5 | 5 | 5 | 4 | 5
Completed | 5 | 5 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 1
Arm/Group | Laminated, Then CJ, Then Infinite, Then Quatro | Laminated, Then CJ, Then Quatro, Then Infinite | Laminated, Then Infinite, Then CJ, Then Quatro | Laminated, Then Infinite, Then Quatro, Then CJ | Laminated, Then Quatro, Then Infinite, Then CJ | Laminated, Then Quatro, Then CJ, Then Infinite
Started | 5 | 5 | 5 | 5 | 4 | 5
Completed | 5 | 5 | 5 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Experimental Socket #1
Arm/Group | Laminated, Then CJ, Then Infinite, Then Quatro | Laminated, Then CJ, Then Quatro, Then Infinite | Laminated, Then Infinite, Then CJ, Then Quatro | Laminated, Then Infinite, Then Quatro, Then CJ | Laminated, Then Quatro, Then Infinite, Then CJ | Laminated, Then Quatro, Then CJ, Then Infinite
Started | 5 | 5 | 5 | 4 | 3 | 5
Completed | 5 | 5 | 5 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash-out 2
Arm/Group | Laminated, Then CJ, Then Infinite, Then Quatro | Laminated, Then CJ, Then Quatro, Then Infinite | Laminated, Then Infinite, Then CJ, Then Quatro | Laminated, Then Infinite, Then Quatro, Then CJ | Laminated, Then Quatro, Then Infinite, Then CJ | Laminated, Then Quatro, Then CJ, Then Infinite
Started | 5 | 5 | 5 | 4 | 3 | 5
Completed | 4 | 5 | 5 | 2 | 3 | 4
Not Completed | 1 | 0 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2 | 0 | 1
Period: Experimental Socket #2
Arm/Group | Laminated, Then CJ, Then Infinite, Then Quatro | Laminated, Then CJ, Then Quatro, Then Infinite | Laminated, Then Infinite, Then CJ, Then Quatro | Laminated, Then Infinite, Then Quatro, Then CJ | Laminated, Then Quatro, Then Infinite, Then CJ | Laminated, Then Quatro, Then CJ, Then Infinite
Started | 4 | 5 | 5 | 2 | 3 | 4
Completed | 4 | 4 | 5 | 2 | 3 | 4
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Wash-out 3
Arm/Group | Laminated, Then CJ, Then Infinite, Then Quatro | Laminated, Then CJ, Then Quatro, Then Infinite | Laminated, Then Infinite, Then CJ, Then Quatro | Laminated, Then Infinite, Then Quatro, Then CJ | Laminated, Then Quatro, Then Infinite, Then CJ | Laminated, Then Quatro, Then CJ, Then Infinite
Started | 4 | 4 | 5 | 2 | 3 | 4
Completed | 3 | 4 | 3 | 2 | 3 | 4
Not Completed | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0 | 0 | 0
Period: Experimental Socket #3
Arm/Group | Laminated, Then CJ, Then Infinite, Then Quatro | Laminated, Then CJ, Then Quatro, Then Infinite | Laminated, Then Infinite, Then CJ, Then Quatro | Laminated, Then Infinite, Then Quatro, Then CJ | Laminated, Then Quatro, Then Infinite, Then CJ | Laminated, Then Quatro, Then CJ, Then Infinite
Started | 3 | 4 | 3 | 2 | 3 | 4
Completed | 3 | 4 | 3 | 2 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This group represents all study participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] — Self reported age in years at time of enrollment
  years | 47.8 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported race and ethnicity
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 28
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 22
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Socket Fit Comfort Score
Description: The Socket Fit Comfort Score (SCS) is a single question in which subjects are asks: "On a scale from 0-10, if 0 represents the most uncomfortable socket fit you can imagine and 10 represents the most comfortable socket fit, how would you score the comfort of the socket fit of your artificial limb at the moment?"
Time Frame: After at least 3 weeks of prosthetic socket use
Population: All participants who successfully wore the socket at home for three weeks are included. We also exclude baseline data from individuals who did not successfully complete at least one experimental socket.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Laminated Socket: During this condition, participants wore their prescribed laminated socket. Three participants were prescribed CJ sockets, rather than laminated and instead were fit with a laminated socket by a study prosthetist for this condition.
- CJ Socket: Participants were fitted with a CJ sail socket (CJ Socket Technologies, Beverly, MA). Three participants were prescribed CJ sails prior to the study initiation.
- Quatro: Participants were fitted with a Quatro socket (Quorum Prosthetics, Windsor, Colorado)
- Infinite Socket: Participant were fitted with an Infinite socket (LiM Innovations, San Francisco, CA)
Arm/Group | Laminated Socket | CJ Socket | Quatro | Infinite Socket
Number analyzed (Participants) | 22 | 16 | 17 | 19
units on a scale | 7.0 (0.5) | 7.4 (0.6) | 7.9 (0.4) | 7.3 (0.5)
Statistical Analysis 1: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; The null hypothesis was that all sockets would have the same SCS; Test type: Superiority; p = 0.553, ANOVA — Statistical significance was set a-priori at p<0.05

2. Primary Outcome: Satisfaction and Quality of Life on the Prosthetic Evaluation Questionnaire (PEQ)
Description: The PEQ consists of 82 items of which 41 items form nine subscales concerning Prosthesis Utility (UT), Residual Limb Health (RL), Appearance (AP), Sounds (SO), Ambulation (AM), Perceived Response (PR), Frustration (FR), Social Burden (SB), and Well-Being (WB). The remaining 41 items are analyzed as single items. These items are scored on a 100-mm visual analog scale with descriptors at the extremes (e.g. never and all the time). The scales are calculated as averages of the items on a metric from 0 to 100 with higher scores indicating better health.
Time Frame: After at least 3 weeks of prosthetic socket use
Population: All participants who successfully completed at least one experimental condition
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Laminated Socket | CJ Socket | Quatro | Infinite Socket
Number analyzed (Participants) | 22 | 16 | 17 | 19
units on a scale
  Frustration Subscale | 54.6 [41.5 to 67.8] | 65.3 [49.6 to 80.9] | 61.7 [46.6 to 76.8] | 51.9 [38.0 to 65.9]
  Perceived Response Subscale | 85.1 [79.5 to 90.8] | 90.0 [83.3 to 96.7] | 89.9 [83.4 to 96.4] | 87.3 [81.3 to 93.3]
  Social Burden Subscale | 70.0 [63.5 to 76.4] | 82.1 [74.4 to 89.8] | 79.8 [72.3 to 87.2] | 77.9 [71.1 to 84.8]
  Ambulation Subscale | 52.4 [45.2 to 59.5] | 66.6 [58.1 to 75.0] | 66.9 [58.7 to 75.0] | 57.1 [49.6 to 64.6]
  Prosthesis Utility Subscale | 59.3 [52.0 to 66.5] | 72.6 [64.0 to 81.2] | 72.2 [63.9 to 83.8] | 62.9 [55.2 to 70.5]
  Residual Limb Health Subscale | 68.4 [62.1 to 74.7] | 71.1 [63.6 to 78.6] | 76.5 [69.3 to 83.8] | 75.9 [69.2 to 82.6]
  Appearance Subscale | 65.3 [58.3 to 72.3] | 76.7 [68.4 to 85.0] | 73.3 [65.3 to 81.3] | 62.1 [54.7 to 69.5]
  Sounds Subscale | 65.2 [55.6 to 74.9] | 78.5 [67.1 to 89.9] | 69.5 [58.4 to 80.5] | 71.0 [61.8 to 82.2]
  Well-Being Subscale | 67.9 [61.7 to 74.1] | 65.4 [58.1 to 72.8] | 77.2 [70.2 to 84.3] | 73.5 [66.9 to 80.1]
Statistical Analysis 1: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; The null hypothesis was that all sockets would be the same; Test type: Superiority — Frustration sub-scale; p = 0.536, ANOVA
Statistical Analysis 2: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority — Perceived Response; p = 0.598, ANOVA
Statistical Analysis 3: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority — Social Burden; p = 0.072, ANOVA
Statistical Analysis 4: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority — Ambulation Sub-scale; p = 0.018, ANOVA
Statistical Analysis 5: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority — Prosthesis Utility; p = 0.037, ANOVA
Statistical Analysis 6: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority — Residual Limb Health; p = 0.254, ANOVA
Statistical Analysis 7: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority — Appearance; p = 0.032, ANOVA
Statistical Analysis 8: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority — Sounds; p = 0.352, ANOVA
Statistical Analysis 9: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority — Well-being; p = .077, ANOVA

3. Primary Outcome: Activities Specific Balance Confidence Scale
Description: The ABC scale is a 16-item self-reported measure scored on a rating scale from 0 to 100, with higher scores indicate greater balance confidence. An average score is calculated by adding all item scores and dividing by the total number of items. The ABC scale has demonstrate high internal consistency, good test-retest validity, and good construct validity in people with lower limb amputation.
Time Frame: After at least 3 weeks of prosthetic socket use
Population: All participants who successfully completed at least one experimental socket are included. One participants surveys for the laminated condition were lost in the mail.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Laminated Socket | CJ Socket | Quatro | Infinite Socket
Number analyzed (Participants) | 21 | 16 | 17 | 19
units on a scale | 68.7 (2.8) | 70.4 (3.3) | 67.8 (3.2) | 68.8 (3.0)
Statistical Analysis 1: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority; p = 0.95, ANOVA; general linear model with socket as fixed factor and participant as random factor

4. Primary Outcome: Mobility as Measured by the 10-meter Walk Test
Description: The 10-m walk test measures elapsed time over 10 m from a standing start. Participants complete one practice trial and then two test trials. The outcome is the average speed walked during the two trials.
Time Frame: after at least 4 weeks of prosthetic socket use
Population: All participants who successfully completed at least one experimental socket were included (n=23). Data is included for all participants who successfully wore the socket home for four weeks before dropping out of the study or failing the socket condition.
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Laminated Socket | CJ Socket | Quatro | Infinite Socket
Number analyzed (Participants) | 22 | 16 | 18 | 16
m/s | 1.06 (.03) | 1.09 (.03) | 1.07 (.03) | 1.08 (.03)
Statistical Analysis 1: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority; p = .853, ANOVA; general linear model with sockets as fixed effect and subjects as random effect

5. Primary Outcome: Mobility as Measured by Timed Up and Go (TUG)
Description: The timed-up-and-go (TUG) assesses several aspects of mobility including getting out of a chair, walking 3 m, turning, and sitting down (Schoppen et al. 1999). The outcome is the time from buttocks off the chair to buttocks down. The best of three trials was recorded.
Time Frame: after at least 4 weeks of prosthetic socket use
Population: All participants who successfully completed at least one experimental socket where included. For those 23 participants, only conditions where the participant wore the socket for four weeks are included
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Laminated Socket | CJ Socket | Quatro | Infinite Socket
Number analyzed (Participants) | 22 | 16 | 15 | 18
seconds | 15.0 (.39) | 14.4 (.48) | 14.4 (.50) | 15.1 (.45)
Statistical Analysis 1: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority; p = 0.565, ANOVA; general linear model with socket as a fixed factor and subjects as a random factor

6. Primary Outcome: Mobility as Measured by Five Times Sit To Stand (FTSTS)
Description: FTSTS is a measure of functional mobility, lower limb strength, and dynamic balance.
Time Frame: after at least 4 weeks of prosthetic socket use
Population: as for outcome 4
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Laminated Socket | CJ Socket | Quatro | Infinite Socket
Number analyzed (Participants) | 22 | 16 | 16 | 18
seconds | 24.9 (1.1) | 21.8 (1.4) | 24.0 (1.4) | 23.9 (1.3)

7. Primary Outcome: Self-reported Mobility Using the Prosthetic Limb Users Survey of Mobility (PLUMS-M) 12-item Short Form
Description: The PLUS-M 12-item short form assess self-reported mobility. The questions are summed and the score is converted to a T-Score (e.g. 50 indicates the population mean with a standard deviation of 10). Values higher than 50 indicate self-reported mobility better than the average person with lower limb amputation, while those less than 50 are below the average.
Time Frame: After at least 3 weeks of prosthetic socket use
Population: All participants who successfully completed at least one experimental socket were included (n=23). Data is included for all participants who successfully wore the socket home for three weeks before dropping out of the study or failing the socket condition. Surveys for one participant in the laminated condition were lost in the mail.
Measure: Mean (Standard Error); unit: T Score
Arm/Group | Laminated Socket | CJ Socket | Quatro | Infinite Socket
Number analyzed (Participants) | 21 | 16 | 17 | 19
T Score | 50.5 (1.0) | 50.6 (1.1) | 52.0 (1.1) | 49.4 (1.0)
Statistical Analysis 1: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority; p = .374, ANOVA; general linear model with socket as fixed factor and subjects as random factor

8. Secondary Outcome: Prosthetic Wear Time
Description: Participants will be given sensors to monitor how many times participants don and doff the prosthesis during the day. This sensor will be attached to each socket after the 3rd week of accommodation. This sensor will be worn for 1 week.
Time Frame: After at least 3 weeks of prosthetic socket use
Population: All participants with data. The data from the sensor was not reliable, so data was used from self report.
Measure: Mean (Standard Deviation); unit: average number of times per day
Arm/Group | Laminated Socket | CJ Socket | Quatro | Infinite Socket
Number analyzed (Participants) | 23 | 16 | 14 | 15
average number of times per day | 1.77 (.837) | 1.49 (1.7) | 1.47 (.53) | 1.05 (.35)

9. Secondary Outcome: Time to Complete the L Test
Description: The L test is a modified version of the TUG which incorporates two transfers and four turns of which at least one would be to the opposite side. The fastest time out of three trials was recorded.
Time Frame: After 4 weeks of prosthetic socket use
Population: as for outcome 4
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Laminated Socket | CJ Socket | Quatro | Infinite Socket
Number analyzed (Participants) | 22 | 16 | 15 | 18
seconds | 33.1 (.8) | 32.2 (1.0) | 31.2 (1.1) | 32.6 (1.0)
Statistical Analysis 1: Comparison: Laminated Socket vs CJ Socket vs Quatro vs Infinite Socket; Test type: Superiority; p = .574, ANOVA; general linear model with socket as a fixed factor and subjects as a random factor

10. Secondary Outcome: Steps Per Day Taken at Home
Description: Participants will wear accelerometers to measure their average step count per day over a one week time frame. Data will be collected after at least three weeks of socket use.
Time Frame: After three weeks of device use
Population: All participants with at least one full day of accelerometer data.
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Laminated Socket | CJ Socket | Quatro | Infinite Socket
Number analyzed (Participants) | 28 | 16 | 15 | 16
steps/day | 2526 (1857) | 2238 (1842) | 2224 (1626) | 2616 (1828)

11. Secondary Outcome: Prosthetic Preference
Description: The prosthetic preference questionnaire consisted of a single question which asked which socket the participant preferred on a 100 mm visual analog scale from their prescribed socket to the test socket. A score of 0 would be 100% preference for their prescribed socket while 100 mm represents 100% preference for the experimental socket.
Time Frame: After at least three weeks of prosthetic socket use.
Population: Data were compared to the participants prescribed socket, which was either laminated (n=26) or CJ (n=3). There is only data for individuals who successfully completed at least two conditions (i.e. baseline and experimental). Since this is a relative measure, there is less data than for other outcomes. For example, only individuals who were prescribed the CJ would have a value for the laminated condition. Several participants also did not complete this survey.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Laminated Socket | CJ Socket | Quatro | Infinite Socket
Number analyzed (Participants) | 1 | 10 | 14 | 13
units on a scale | 4 (NA) — There is only one data point so a standard error cannot be calculated | 33.4 (11.6) | 48.3 (11.0) | 37.4 (9.6)

ADVERSE EVENTS:
Time Frame: over 4 weeks of prosthetic socket use, up to two months
Arm/Group | Laminated Socket | CJ Socket | Quatro | Infinite Socket
All-Cause Mortality (participants affected / at risk) | 1/28 | 0/25 | 0/20 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/25 | 1/20 | 1/24
Other Adverse Events (participants affected / at risk) | 2/28 | 13/25 | 7/20 | 10/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laminated Socket (N=28) | CJ Socket (N=25) | Quatro (N=20) | Infinite Socket (N=24)
Death (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Physician reported that participant passed away. They were not in an experimental socket at the time as the study was on a pause for COVID-19. Cause of death is not known but a choice of organ system was made as there is no unknown category.
Cancer (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The participant experienced a reoccurrence of cancer so they dropped out of the study for treatment.
Hospitalization (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The participant experienced excessive swelling of their residual limb and was hospitalized. They had already been fit with the Infinite check socket but had not received the definitive and therefore was wearing their prescribed socket at the time.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laminated Socket (N=28) | CJ Socket (N=25) | Quatro (N=20) | Infinite Socket (N=24)
Wound (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 3 (3) — Participant developed a wound on their residual limb
Injurious fall requiring medical attention (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) — Participant experienced an injurious fall that resulted in them seeking medical attention
Instability/Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (9) | 2 (2) | 5 (5) — Participant experienced limb instability or discomfort that limited or prevented them from wearing the socket
Device Issues (Product Issues) | 0 (0) | 0 (0) | 4 (4) | 1 (1) — Participant reported experiencing issues with the socket such as loss of suspension, part of the socket breaking off, issues with components, etc.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT04038580/Prot_SAP_000.pdf